CLINICAL TRIAL: NCT05554055
Title: Correlation Between LR-ACT and Anti Xa Activity During Endovascular Surgery Procedures.
Brief Title: Correlation Between LR-ACT and Anti Xa Activity During Endovascular Surgery Procedures. AXAES (Anti Xa vs ACT-LR in Endovascular Surgery)
Acronym: AXAES
Status: Withdrawn | Type: Observational
Why Stopped: The AXAES study was stopped mainly for logistical and organizational reasons. The machine needed to carry out the examinations was no longer available, making it impossible to continue the study.
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0104
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Aortic Diseases; Arterial Disease; Thrombosis
Keywords: Complex aortic endovascular repair; Arterial recanalization; Deep veinous recanalization; Anti Xa; LR-ACT; Heparin; Endovascular procedures
MeSH Terms: conditions — Aortic Diseases; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Anti Xa activity measurement. — Arterial blood samples of 3cc will be taken during the procedure at each ACT. Blood samples will be sent to the lab for anti Xa activity measurement.

SUMMARY:
Activated clotting time (ACT) is currently recommended to monitor high concentrations heparin anticoagulation. ACT-LR was specifically designed to measure the activity of low dose of heparin used during endovascular surgery. The correlation between ACT-LR and Anti Xa activity which is considered as the gold standard seems to be debated.

Few studies in literature had shown controversial results. These studies were conducted in patients who underwent open as endovascular surgery. However, the ACT monitoring is not recommended in open surgery. In addition, heparin administration protocols are not described and specific to each centre.

In this study investigators want to study the correlation between LR-ACT and anti Xa after introducing a heparin protocol during complex endovascular procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 ans
* Weight ≥ 37,5 kg
* Patients operated for
* complex endovascular aortic aneurysm repair
* deep vein recanalization
* complex arterial revascularization (TASC D lesions)
* Patient informed of the study details and who didn't opposed to participate in this research

Exclusion Criteria:

* Known allergy to heparin
* Known hepatic insufficiency with repercussion on coagulation
* Thrombocytopenia
* Known hemostasis disorders
* Anemia defined HB<8 g/L
* Pregnant women
* Persons deprived of their liberty by a judicial or administrative decision
* Persons subject to psychiatric care
* Persons admitted to a health or social establishment for purposes other than research
* Adults subject to a legal protection measure (guardianship, curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who will undergo an endovascular surgery in the centre.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Correlation between ACT (second) realized in operative room and Anti Xa activity (UI/ml) results provide by the lab. | During surgery - 1 day
  Following the heparin administration protocol, each ACT measurement will be associated to a blood samples for anti Xa activity measurement.
  Retrospectively, anti Xa results will be analyze and compare to ACT value which will be report in the operative report.
  The blood samples will be taken in operative room during endovascular procedures as defined in the protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de chirurgie vasculaire (U50) Hôpital Louis Pradel - HCL, Bron, France

IPD SHARING:
Plan to Share IPD: No